CLINICAL TRIAL: NCT04120012
Title: The Effect of Frailty to Intraoperative Hemodynamic Instability and Perioperative Complications in the Elderly: a Prospective Observational Study
Brief Title: The Effect of Frailty to Perioperative Complications in the Elderly
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-8-20
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2022-05

CONDITIONS: Fragility; Intraoperative Hypotension; Perioperative Complication
Keywords: Frailty; Intraoperative Hypotension; Perioperative Complication; Elderly
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and urine samples will be collected from patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
With the progression of population aging, the number of elderly patients undergoing surgery is increasing as well. However, as the condition of health differs greatly between individual elderly patients even of the same age, it is a necessity to evaluate elderly patients thoroughly and individually for better management of perioperative care.

Frailty is a condition in which patients are impaired at physical reserve and homeostatic control. Frail elderly people are at higher risk of morbidity and mortality after exposure to a stressor. Frail patients are at higher risk of perioperative complications and longer hospital stay. However, there has been no standard criteria or tool to evaluate frailty in the elderly. Neither has there been enough evidence explaining the mechanism between frailty and increased perioperative complications. Therefore, in this study we aim to discover the relationship between frailty and intraoperative hemodynamic instability, as well as perioperative complications in the elderly patients, hoping to find an adequate and practical model for preoperative assessment in the elderly hopefully for better perioperative outcome.

ELIGIBILITY:
Inclusion Criteria:

* age≥65 years
* elective major non-cardiac surgery
* general anesthesia
* American Society of Anesthesiologists(ASA) grade I,II,III
* study protocol fully understood by the patients, written consent obtained

Exclusion Criteria:

* emergency surgery
* in active state of infection or inflammation
* chronic kidney disease(CKD) stage 5
* having conditions that would interfere accurate measurement of upper extremity blood pressure (e.g. subclavian artery stenosis)
* having conditions that would interfere assessment of frailty assessment (e.g. mental disorder, hearing disorder)
* study protocol not fully understood, no written consent obtained

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study intend to include elderly patients (≥65years) who undergoes elective major non-cardiac surgery who can cooperate with upper extremity blood pressure measurement and frailty assessment.
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative hypotension | Intraoperative
  Intraoperative hypotension includes post induction hypotension(PIH), early intraoperative hypotension(eIOH) and late intraoperative hypotension(lIOH). Hypotension is defined as a systolic blood pressure less than 90mmHg or a relative decrease more than 30% compared to baseline blood pressure, or mean arterial pressure less than 65mmHg or a decrease more than 30% compared to baseline. PIH is defined as a hypotension within 20 minutes after anesthesia induction, or before surgical incision. eIOH is defined as hypotension within 30 minutes after the start of surgery. lIOH is defined as hypotension that happen 30 minutes after the start of surgery until the end of surgery.
Incidence of intraoperative hemodynamic instability | Intraoperative
  Intraoperative hemodynamic instability is defined as a definite change of systolic blood pressure, or mean arterial pressure, or diastolic pressure, or pulse pressure more than 15% or the need for vasoactive agents.

SECONDARY OUTCOMES:
Incidence of postoperative complications | Within 30days after surgery
  Postoperative complications will be recorded according to medical records and laboratory results within 30 days after surgery according to Clavien-Dindo classification of surgical complications. Incidence of each grade will be calculated as outcome. Postoperative acute kidney injury will be assessed by analysis of urinary and serum biomarkers before and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Li Xu, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China